CLINICAL TRIAL: NCT07136766
Title: An 18 Week Study to Assess the Efficacy of a Test Product Used in Combination With a Currently Marketed Prescription Product
Brief Title: An 18-week Study to Evaluate a Test Product With a Marketed Prescription Product
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Good Molecules, LLC (Industry)
Collaborators: Validated Claim Support (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS251008
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Product (Experimental)
  Interventions: Drug: Facial Toner
- Control Product (Sham Comparator)
  Interventions: Other: Placebo Toner

INTERVENTIONS:
Drug: Facial Toner — Brightening Toner
  Arms: Test Product
Other: Placebo Toner — Placebo Control Toner
  Arms: Control Product

SUMMARY:
The purpose of this study is to assess the efficacy (ability to produce a desired or intended result) of a topical product (applied to the skin) to improve skin lightness, skin condition and appearance (hyperpigmentation [dark spots], brightness/radiance [healthy vibrant appearance], skin texture [smoothness]) on ] the face over a period of eighteen (18) weeks. The data collected may support the company in developing marketing claims for its product.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with facial hyperpigmentation and/or melasma.
2. Individuals willing to use a generic 4% Hydroquinone prescription topical cream up to 10 weeks for the duration of the study.
3. Individuals willing to refrain from use of other drugs or skincare intended to treat hyperpigmentation, other than study-specific products (prescription drug, test product, SPF 50) for the duration of the study.
4. Individuals who are able to cooperate with the Principal Investigator and study personnel throughout the duration of the study and are willing to comply with all study procedures, methods, evaluations, and study product use.
5. Individuals who are able to read, understand and willing to sign an informed consent for this specific study and have completed all site required documentation prior to study enrollment (Registration and Medical History).
6. Individuals who are able to receive emails on their cellular phones and are capable of completing electronic Informed Consents, Photo Model Releases, and/or Questionnaires on their device.
7. Individuals willing to be photographed and sign a model release.

Exclusion Criteria:

1. Individuals with known allergies and/or reactions to Hydroquinone.
2. Individuals currently participating in other clinical studies that are testing a face product.
3. Individuals with uncontrolled medical condition(s), including dermatological problems, which could put them at risk in the opinion of the Principal Investigator or compromise the study outcome and/or chronic or serious diseases and conditions which would prevent participation in this clinical study such as cancer, AIDS, insulin-dependent diabetes, renal impairment, mental illness, and/or drug/alcohol addiction.
4. Individuals with a history of melanoma, or a treated skin cancer within the last 5 years.
5. Individuals who are pregnant, lactating, or planning to become pregnant. Individuals who become pregnant during the study must inform the Principal Investigator immediately.
6. Individuals who are unreliable or unlikely to be available for the duration of the study.
7. Individuals with a history of allergic reactions, skin sensitization and/or known allergies to cosmetic and personal care products/ingredients.
8. Individuals who are immunocompromised.
9. Individuals who are employees of VCS, other testing firms/laboratories, consumer product, and/or raw goods manufacturers/suppliers.
10. Individuals who are unable to communicate or cooperate with the Principal Investigator/study personnel due to language problems, poor mental development, or impaired cerebral function.
11. Individuals who started hormones within the last three months preceding the commencement of the study.
12. Individuals who are using oral contraception for less than three months before study commencement or who have changed their contraceptive method within the three months before the Baseline visit or planning to modify their contraception treatment within the duration of the study.
13. Individuals who have regular salon and/or dermatological procedures that can interfere with study results (Microdermabrasion, Fillers, Facial Peels, etc.) and are not willing to stop throughout the study.
14. Individuals with facial tattoos and facial piercings (that can't be removed).
15. Individuals with tattooed/permanent make up (i.e., eyeliner, eyebrows, lip liner, etc.), eyebrow microblading, and/or eyelash extensions.
16. Individuals who plan to change their hairstyle throughout the course of the study or who wear hair coverings regularly (i.e., wigs, coloring, extensions, etc.).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Skin Lightness | 18 weeks
  L* and Individual Typology Angle

SECONDARY OUTCOMES:
Facial Hyperpigmentation | 18 weeks
  Analyzed by Expert Grading in a 10-point ordinal scale (0 = positive anchor of uniform, even appearance, and 9 = negative anchor of uneven, discolored, pigmentation present)
Facial Skin Texture | 18 weeks
  Analyzed by Expert Grading in a 10-point ordinal scale (0 = positive anchor of smooth, even surface appearance, and 9 = negative anchor of rough, uneven surface appearance)
Facial Brightness/Radiance | 18 weeks
  Analyzed by Expert Grading in a 10-point ordinal scale (0 = positive anchor of radiant, glowing appearance, and 9 = negative anchor of dull/lackluster)
Volunteer's opinion on product | 18 weeks
  Subjective Questionnaire
Facial skin changes via images | 18 weeks
  Photo analysis acquired via Visia CR Imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Validated Claim Support, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumann L. Skin ageing and its treatment. J Pathol. 2007 Jan;211(2):241-51. doi: 10.1002/path.2098. PMID 17200942
- [Background] Samson N, Fink B, Matts PJ. Visible skin condition and perception of human facial appearance. Int J Cosmet Sci. 2010 Jun;32(3):167-84. doi: 10.1111/j.1468-2494.2009.00535.x. Epub 2009 Nov 3. PMID 19889046

DOCUMENTS (1):
  • Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT07136766/ICF_000.pdf